CLINICAL TRIAL: NCT00525291
Title: Prospective, Randomized Multicenter Study to Assess the Outcome of Conservative 3T Treatment With EMG-Biofeedback
Brief Title: Triple Target Treatment (3T) Which Combines Stimulation With Amplitude Modulated Middle Frequency (AM-MF), Electromyography (EMG)-Triggered Stimulation and EMG-Biofeedback Compared With EMG-Biofeedback in Anal Incontinence
Acronym: 3T-AI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Giessen (Other)
Responsible Party: Universitätsklinikum Gießen und Marburg, Standort Gießen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 83/07 ethics comm. Giessen
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-01

CONDITIONS: Fecal Incontinence
Keywords: Exercise Therapy; Biofeedback (Psychology); Adult; Fecal Incontinence/*therapy; EMG - Biofeedback; EMG - Triggered Stimulation; Augmented biofeedback
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EMG-biofeedback plus EMG-triggered AM-MF-stimulation (Experimental)
  Interventions: Device: Combination of EMG-biofeedback plus EMG-triggered AM-MF-stimulation
- EMG-biofeedback alone (Active Comparator)
  Interventions: Device: EMG-biofeedback alone

INTERVENTIONS:
Device: Combination of EMG-biofeedback plus EMG-triggered AM-MF-stimulation — In the 3T arm, patients were stimulated with a carrier wave of 25 KHz and biphasic modulations of the pulse train of 40 Hz. Anxious patients trained at first only in the biofeedback mode. The stimulation was introduced after four weeks for these patients. Patients were instructed to carry out the training at home, with an alternating combination in the morning and with EMG-triggered stimulation in the evening, each for 20-minute periods. Apart from this, the protocol of the active treatment group was identical to that of the control group.
  Arms: EMG-biofeedback plus EMG-triggered AM-MF-stimulation
Device: EMG-biofeedback alone — In the biofeedback arm, patients were instructed to carry out EMG-biofeedback training at home, standing, mornings and evenings, for 20-minute periods. The core of the task was to pull the plug-electrode upward inside the anal channel, like a lift, and to hold it there during varying periods of tension. This can only be done successfully if the perineum rises and at the same time the puborectal muscle is activated. Just squeezing the sphincter muscles does not produce this lifting effect.
  Arms: EMG-biofeedback alone

SUMMARY:
The efficacy of biofeedback and/or low frequency electrical stimulation for the treatment of anal incontinence has not been proven. First, large well-designed clinical trials are missing. Second, only few patients reach therapeutically relevant intensities with low frequency stimulation. In this study, a novel therapeutic concept, termed triple target treatment (3T) was evaluated. 3T combines stimulation with amplitude modulated middle frequency (AM-MF), electromyography (EMG)-triggered stimulation and EMG-biofeedback. 3T was compared with EMG-biofeedback alone after a nine month treatment period.

Methods In this parallel-group randomised multicenter study with blinded observer we enrolled 158 patients with anal incontinence. Primary endpoints were changes from baseline to nine months in the Cleveland Clinic Score (CCS) and the St. Mark's score (Vaizey score).

ELIGIBILITY:
Inclusion Criteria:

* All Patients with fecal incontinence I-III.

Exclusion Criteria:

* All Patients with CID´s
* Definite or possible pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Cleveland Clinic Incontinence Score (CCS) in its validated German form after nine months, compared to baseline | 9 months after randomization
Validated new St. Mark's incontinence score (Vaizey score) in its adapted German form after nine months, compared to baseline. | 9 months after randomization

SECONDARY OUTCOMES:
CCS score after six or three months, compared to baseline | 3 months, 6 months after randomization
Adapted Vaizey score after six or three months compared to baseline | 3 months, 6 months
Quality of life according to the Fecal Incontinence Quality of Life Scale (FIQoL) in its validated German form after nine months compared to baseline, as well as between the two treatment groups over the course of time as compared to baseline | 9 months after randomization
Track record of the treatment: 1. Continent, 2. Grade improvement (grade II or III to grade I), 3. Frequency improvement: (same grade, >= 2 points improvement in CCS), 4. no improvement, or deterioration, 5. early dropouts. | 9 months after randomization
Use of stool regulating medication. Specifically, if biofeedback and 3T increase continence, the use of any stool regulating medication (Fleawort seeds, Loperamide, teas, etc.) should decrease in the course of the trial. | 9 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Thilo Schwandner, Dr., Principal Investigator — University of Giessen
Locations (1):
- University of Gießen, Dept. of General Surgery, Giessen, Hesse, Germany

REFERENCES:
- [Derived] Schwandner T, Heimerl T, Konig IR, Kierer W, Roblick M, Bouchard R, Unglaube T, Holch P, Kolbert G, Padberg W, Ziegler A. [3T-AI: a new treatment algorithm for anal incontinence with a higher evidence level]. Zentralbl Chir. 2012 Aug;137(4):345-51. doi: 10.1055/s-0031-1271468. Epub 2011 Sep 27. German. PMID 21968596
- [Derived] Schwandner T, Konig IR, Heimerl T, Kierer W, Roblick M, Bouchard R, Unglaube T, Holch P, Ziegler A, Kolbert G. Triple target treatment (3T) is more effective than biofeedback alone for anal incontinence: the 3T-AI study. Dis Colon Rectum. 2010 Jul;53(7):1007-16. doi: 10.1007/DCR.0b013e3181db7738. PMID 20551752